CLINICAL TRIAL: NCT06488001
Title: Preoperative Use of Pantoprazole for Prevention of Post Operative Nausea and Vomiting in Gynecologic Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NMCP.2021.0131
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; Postoperative nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Pantoprazole; Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): This arm receives the placebo drug. This medication is taken the night before, 2 hours before surgery, and the night after surgery.
  Interventions: Drug: Placebo
- Active (Active Comparator): This arm receives the pantoprazole 40mg tablet. This medication is taken the night before, 2 hours before surgery, and the night after surgery.
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: pantoprazole — Pantoprazole 40mg given the night before surgery, 2 hours prior to surgery, and the evening after surgery.
  Other Names: proton pump inhibitor
  Arms: Active
Drug: Placebo — Placebo given the night before surgery, 2 hours prior to surgery, and the evening after surgery.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to see if pantoprazole (a proton pump inhibitor used for acid reflux/heart burn) can reduce nausea and vomiting after gynecologic surgery in women between the ages of 18 and 79.

Researchers will compare a placebo to the active medication.

Participants will be asked to take three pills around their surgery, two taken before and one taken the night after.

DETAILED DESCRIPTION:
Randomization Recruited subjects will be randomly assigned a study number and be provided a numerically matching medication packet prepared in advance by pharmacy support staff. Identical opaque gelatin capsules will be prepared in advance containing either placebo or 40 mg of Pantoprazole, each medication packet will have three capsules of either active drug or placebo. The patient and all study members will be blinded. Participants will be instructed when to take their specific medication (PPI or placebo) prior to surgery along with their other ERAS protocol instructions.

Study Medication/Placebo Administration Subjects will take either oral Pantoprazole 40 mg or placebo the evening prior to surgery, 2 hours prior to scheduled surgery (time to peak bioavailability is 2.5 hrs in adults) and 12 hours following surgery completion. The final dose is to provide additional effect given that PONV can continue up to 24 hours following surgery. All surgeries at this facility utilize an ERAS protocol includes the perioperative use of Zofran 4 mg and Decadron 4 mg for all patients; this practice will continue unchanged for participating patients.

Data Collection/Post-Operative Patient Satisfaction Evaluation Subjects will be evaluated postoperatively with a visual analog scale (VAS) to determine incidence and severity of PONV; this has been used similarly in prior studies. A score of 0 indicates no nausea and higher scores reflect progressively greater severity. Assessment with VAS will be conducted two hours after and the morning following surgery completion; scores will be compared between groups. The VAS will be administered in person by study personnel while patients remain in hospital. Study personnel will administer the VAS by phone for patients who have been discharged by the morning following surgery. Time to first meal (PO) will also be measured and compared as will the use of rescue antiemetics to treat nausea postoperatively. Patients will also have a postoperative telehealth visit one week following their operation to review patient satisfaction and rate their experience using the Treatment Acceptability and Preference (TRAP) Questionnaire. This is a validated standard questionnaire that will be verbally administered by study personnel and used to assess patient satisfaction with their perioperative treatment specific to PONV [14]. All data will be collected and stored on password protected excel spreadsheets or in a locked secure environment in the Women's Health Clinic. Subject ID log will be kept separate from data collection tool to maintain blinding by a study team member. Essentris records will be reviewed by the study team member to specifically evaluate time to first meal, reported vomiting and any rescue antiemetic use. All data collected to include VAS and TRAP scores will be collected and stored on password protected excel spreadsheets. Subject ID log will be kept separate from data collection tool to maintain blinding. Analysis will be conducted on appropriate statistical software. To confirm accurate data entry from Essentris, 10% of patient records will be randomly reviewed by a second study investigator (other than the original study team member) and compared prior to data analysis. If any discrepancies are identified in this process, Essentris data will then be reviewed again for all study participants. A list of all discrepancies will be maintained and adjudicated by a third investigator to verify accuracy.

Incidental Malignancy If an unexpected malignancy is found during the surgical procedure, the subject will be withdrawn from the study and all data collected prior to surgery will be discarded.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective gynecological surgery by either an open abdominal or minimally invasive approach (to include both endoscopic and vaginal). Procedure must be performed under general anesthesia.

Exclusion Criteria:

* Pregnant,
* Patients with gastrointestinal disease requiring ongoing medical management.
* Prior gastrointestinal surgery with the exception of diagnostic procedures, appendectomy and cholecystectomy.
* Patients with a history of H2 receptor blocker use, proton pump inhibitor use or other GERD specific therapy within 30 days of surgery.
* Any patient identified by their surgical care team as having a history of PONV warranting additional perioperative prophylaxis.
* Known r suspected malignancy
* Lactose intolerance

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Nausea and Vomiting | From enrollment until their postoperative visit at 6 weeks
  Postoperative nausea and vomiting compared between two groups using Visual Analog Scale from 0-10. A score of 0 indicates no nausea and higher scores reflect progressively greater severity.

SECONDARY OUTCOMES:
Time to Oral Intake | From surgery until first meal, usually within a few hours.
  Measure the time from surgery until patients can tolerate oral intake.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Timmerman, DO, Principal Investigator — United States Naval Medical Center, Portsmouth
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fortier J, Chung F, Su J. Unanticipated admission after ambulatory surgery--a prospective study. Can J Anaesth. 1998 Jul;45(7):612-9. doi: 10.1007/BF03012088. PMID 9717590
- [Background] Sidani S, Epstein DR, Bootzin RR, Moritz P, Miranda J. Assessment of preferences for treatment: validation of a measure. Res Nurs Health. 2009 Aug;32(4):419-31. doi: 10.1002/nur.20329. PMID 19434647
- [Background] Boogaerts JG, Vanacker E, Seidel L, Albert A, Bardiau FM. Assessment of postoperative nausea using a visual analogue scale. Acta Anaesthesiol Scand. 2000 Apr;44(4):470-4. doi: 10.1034/j.1399-6576.2000.440420.x. PMID 10757584
- [Background] Apfel CC, Roewer N, Korttila K. How to study postoperative nausea and vomiting. Acta Anaesthesiol Scand. 2002 Sep;46(8):921-8. doi: 10.1034/j.1399-6576.2002.460801.x. PMID 12190791
- [Background] Nebel OT, Fornes MF, Castell DO. Symptomatic gastroesophageal reflux: incidence and precipitating factors. Am J Dig Dis. 1976 Nov;21(11):953-6. doi: 10.1007/BF01071906. PMID 984016
- [Background] Kwon YS, Choi JW, Lee HS, Kim JH, Kim Y, Lee JJ. Effect of a Preoperative Proton Pump Inhibitor and Gastroesophageal Reflux Disease on Postoperative Nausea and Vomiting. J Clin Med. 2020 Mar 18;9(3):825. doi: 10.3390/jcm9030825. PMID 32197451
- [Background] Koivuranta M, Laara E, Snare L, Alahuhta S. A survey of postoperative nausea and vomiting. Anaesthesia. 1997 May;52(5):443-9. doi: 10.1111/j.1365-2044.1997.117-az0113.x. PMID 9165963
- [Background] Apfel CC, Heidrich FM, Jukar-Rao S, Jalota L, Hornuss C, Whelan RP, Zhang K, Cakmakkaya OS. Evidence-based analysis of risk factors for postoperative nausea and vomiting. Br J Anaesth. 2012 Nov;109(5):742-53. doi: 10.1093/bja/aes276. Epub 2012 Oct 3. PMID 23035051
- [Background] Apfel CC, Turan A, Souza K, Pergolizzi J, Hornuss C. Intravenous acetaminophen reduces postoperative nausea and vomiting: a systematic review and meta-analysis. Pain. 2013 May;154(5):677-689. doi: 10.1016/j.pain.2012.12.025. Epub 2013 Jan 11. PMID 23433945
- [Background] Apfel CC, Kranke P, Eberhart LH, Roos A, Roewer N. Comparison of predictive models for postoperative nausea and vomiting. Br J Anaesth. 2002 Feb;88(2):234-40. doi: 10.1093/bja/88.2.234. PMID 11883387
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Carlisle JB, Stevenson CA. Drugs for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD004125. doi: 10.1002/14651858.CD004125.pub2. PMID 16856030
- [Background] Kalogera E, Dowdy SC. Enhanced Recovery Pathway in Gynecologic Surgery: Improving Outcomes Through Evidence-Based Medicine. Obstet Gynecol Clin North Am. 2016 Sep;43(3):551-73. doi: 10.1016/j.ogc.2016.04.006. PMID 27521884
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299